CLINICAL TRIAL: NCT00180830
Title: Open Label, Pilot Phase II Study of Glivec in Children and Adolescents With Life Threatening Diseases Known to Be Associated With One or More Glivec-Sensitive Tyrosine Kinases
Brief Title: Glivec Phase II Pediatric Study
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EGPS-01; CSET-2002/940; CSTI 571BFR10
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2006-09-11 (Estimated); Status verified 2006-09

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Imatinib Mesylate

INTERVENTIONS:
Drug: Glivec
Drug: Gleevec

SUMMARY:
The purpose of this study is to determine whether Glivec is effective, in children, adolescents and young adults, in the treatment of malignant disease in which evidence suggests a potential pathogenic role of one or more of the tyrosine kinases known to be inhibited by Glivec.

ELIGIBILITY:
Inclusion Criteria:

* Patients from 6 months to 21 years of age.
* Malignant disease documented by conventional criteria to be refractory to standard, approved therapy, or for which no conventional therapies of definitive benefit exist.
* Immunohistochemistry documentation of positivity of either Kit (CD117) or PDGF-R in tumor tissue relevant. Each positive tumor will be centrally reviewed before inclusion of the patient in the trial.
* Measurable or evaluable disease.
* WHO Performance status 0,1, or 2 or Lansky Play Scale >= 50%.
* Adequate organ function, defined as the following: total bilirubin < 1.5 x ULN, SGOT and SGPT < 2.5 x UNL (or < 5 x ULN if hepatic disease involvement is present), creatinine < 1.5 x ULN, ANC > 1x 109/L, platelets > 75 x 109/L.
* Female patients of child-bearing potential must have negative pregnancy test within 7 days before initiation of study drug dosing.
* Male and female patients of reproductive potential must agree to employ an effective barrier method of birth control throughout the study and for up to 3 months following discontinuation of study drug.
* Life expectancy of more than 6 weeks.
* Written, voluntary, informed consent, including consent for retrieval and investigational use of tissue samples for evaluation signed by parents or young adult patients.
* National and, when needed, local ethical approval.

Exclusion Criteria:

* Patient with hematological disease positive for the chimeric BCR-ABL fusion protein or for c-kit.
* Patient has received any other investigational agents within 28 days of first day of study drug dosing.
* Female patients who are pregnant or breast-feeding.
* Patient has another severe and/or life-threatening medical diseasePatient has an acute or known chronic liver disease (e.g., chronic active hepatitis, cirrhosis).
* Patient has a known diagnosis of human immunodeficiency virus (HIV) infection.
* Patient has received chemotherapy within 4 weeks (6 weeks for nitrosourea, mitomycin-C or any antibody therapy) prior to study entry unless urgent enrollment needed and approved by the study coordinator.

Ages: 6 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36
Dates: Start 2003-12

PRIMARY OUTCOMES:
- Tumour Response

SECONDARY OUTCOMES:
Progression-free Survival, overall Survival, safety and tolerability, pharmacokinetic profile and pharmacodynamics of Glivec, pharmacogenetics

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Vassal, MD,PhD, Study Chair — Gustave Roussy, Cancer Campus, Grand Paris; Bruce Morland, Study Chair — Birmingham Children's Hospital
Locations (3):
- Institut Gustave-Roussy, Villejuif, France
- Emma Kinderziekenhuis AMC, Amsterdam, Netherlands
- Birmingham Children's Hospital, Birmingham, United Kingdom